CLINICAL TRIAL: NCT05118802
Title: Measuring the Impact of MANNA s Medically Tailored Meal Program in Patients With a Non-terminal Cancer Diagnosis
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 21G.671; JT 17820 (Other: JeffTrial Number); 080 - 31050 - E269 (Other Grant/Funding Number: MANNA Institute)
Record Dates: First submitted 2021-09-21; First posted 2021-11-12 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (interview, survey): Part I: Patients and clinicians attend semi-structured interviews over 20-30 minutes or cognitive interviews over 60 minutes in support of survey refinement.
  Part II: Patients complete survey over 15 minutes.
  Interventions: Other: Interview; Other: Survey Administration

INTERVENTIONS:
Other: Interview — Attends Interviews
Other: Survey Administration — Complete Survey

SUMMARY:
This study identifies patient-important outcome measures and develops a survey that assesses the impact of nutritional interventions among cancer patients. Currently, data on the impact of medically tailored meals on outcomes that are meaningful to patients, providers, and payers are limited. For this reason, access to medically tailored meals as a covered benefit for cancer patients is limited. Thus, there is a need to explore the efficacy of nutritional interventions among this population. This study identifies outcome measures for nutritional interventions that are meaningful to patients and providers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify patient-important outcomes related to receiving nutrition services by engaging patients with cancer and clinicians.

II. To conduct cognitive interviews to assess comprehension, acceptability, and appropriateness of patient-identified outcomes in aim 1.

III. To pilot test the use of the nutrition-related outcome measures identified in aim 1 among a sample of oncology patients.

OUTLINE:

Part I: Patients and clinicians attend semi-structured interviews over 20-30 minutes or cognitive interviews over 60 minutes in support of survey refinement.

Part II: Patients complete survey over 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1 PATIENTS: SKCC oncology patients
* AIM 1 PATIENTS: Currently receiving cancer treatment
* AIM 1 PATIENTS: 18 years or older
* AIM 1 PATIENTS: English speaking

  * Pending funding and staff abilities, efforts will be made to include other languages if possible
* AIM 1 PATIENTS: 10 patients have received MANNA services in past 6 months
* AIM 1 PATIENTS: 10 patients currently receiving cancer treatment for curative intent, screen positive for nutrition risk, and report food insecurity

  * Nutrition risk = a score of >= 2 on the Malnutrition Screening Tool, weight loss of 5% over 1 months, or weight loss of > 10% over 6 months
* AIM 1 PATIENTS: 10 patients currently receiving cancer treatment for curative intent, screen positive for nutrition risk, and do not report food insecurity
* AIM 1 CLINICIANS: Providing care/support for oncology patients
* AIM 1 CLINICIANS: English speaking
* AIM 2 PATIENTS: Current SKCC oncology patient
* AIM 2 PATIENTS: 18 years or older
* AIM 2 PATIENTS: English speaking

  * Pending funding and staff abilities, efforts will be made to include other languages if possible
* AIM 2 PATIENTS: 3-5 patients have received MANNA services in past 6 months
* AIM 2 PATIENTS: 3-5 patients currently receiving cancer treatment for curative intent, screen positive for nutrition risk, and report food insecurity

  * Nutrition risk = a score of >= 2 on the Malnutrition Screening Tool, weight loss > 5% over 1 month, or weight loss of > 10% over 6 months
* AIM 2 PATIENTS: 3-5 patients currently receiving cancer treatment for curative intent, screen positive for nutrition risk, and do not report food insecurity
* AIM 3 SKCC PATIENTS: Receiving active cancer treatment for curative intent
* AIM 3 SKCC PATIENTS: Meet MANNA eligibility criteria
* AIM 3 SKCC PATIENTS: Have a phone number or email address for contacting
* AIM 3 SKCC PATIENTS: 18 years or older *Pending funding and staff abilities, efforts will be made to include other languages if possible
* AIM 3 MANNA CLIENTS: Have any cancer diagnosis
* AIM 3 MANNA CLIENTS: Currently receiving MANNA meals
* AIM 3 MANNA CLIENTS: Have a phone number or email address for contacting
* AIM 3 MANNA CLIENTS: 18 years or older
* AIM 3 MANNA CLIENTS: English speaking * Pending funding and staff abilities, efforts will be made to include other languages if possible

Exclusion Criteria:

* AIM 1 PATIENTS: Unable to provide consent (as assessed by team member conducting enrollment, with use of teachback)
* AIM 1 PATIENTS: Lives in a facility that provides nutrition services (e.g., nursing home, rehab facility, incarcerated, emergency shelter)
* AIM 1 PATIENTS: Homelessness
* AIM 1 CLINICIANS: Unable to provide consent (as assessed by team member conducting enrollment, with use of teachback)
* AIM 2 PATIENTS: Unable to provide consent (as assessed by team member conducting enrollment, with use of teachback)
* AIM 2 PATIENTS: Lives in a facility that provides nutrition services (e.g., nursing home, rehab facility, incarcerated, emergency shelter)
* AIM 2 PATIENTS: Homelessness
* AIM 3 SKCC PATIENTS: Unable to provide consent (as assessed by team member conducting enrollment, with use of teachback)
* AIM 3 SKCC PATIENTS: Lives in a facility that provides nutrition services (e.g., nursing home, rehab facility, incarcerated, emergency shelter)
* AIM 3 SKCC PATIENTS: Homelessness
* AIM 3 MANNA CLIENTS: Unable to provide consent (as assessed by team members conducting enrollment, with use of teachback)
* AIM 3 MANNA CLIENTS: Homelessness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population includes cancer patients at Sidney Kimmel Cancer Center (SKCC), clinicians and MANNA clients.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
identify patient-important outcomes related to receiving nutrition services by engaging patients with cancer and clinicians | At study completion; approximately 60 minutes
  Reported as average time required to complete each assessment.
Usability | At study completion; approximately 60 minutes
  Reported as average time required to complete each assessment.
Feasibility | At study completion; approximately 60 minutes
  Reported as the number of participants who are able to complete the entire list of assessments to receive nutrition services.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States